CLINICAL TRIAL: NCT05746143
Title: The Effect of Zolpidem on Outcomes Following Lumbar Spine Fusion: A Randomized Control Trial
Brief Title: The Effect of Zolpidem on Outcomes Following Lumbar Spine Fusion
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Raymond Hah, Assistant Professor of Clinical Orthopaedic Surgery, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HS-22-00529
Record Dates: First submitted 2023-02-07; First posted 2023-02-27 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Spine Fusion; Lumbar Spine Degeneration; Pain, Postoperative; Lumbar Spine Spondylosis
Keywords: Lumbar Spine Fusion; Zolpidem; Postoperative Outcomes
MeSH Terms: conditions — Pain, Postoperative | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zolpidem (Experimental)
  Interventions: Drug: Zolpidem Tartrate 10 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zolpidem Tartrate 10 mg — two days preoperatively and five days postoperatively
  Arms: Zolpidem
Drug: Placebo — two days preoperatively and five days postoperatively
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate if peri-operative zolpidem for posterior lumbar spinal fusion improves patient reported outcomes following surgery.

DETAILED DESCRIPTION:
Patients who are undergoing one- to three-level spinal fusion for degenerative lumbar disease will be recruited. They will be randomized to either receive zolpidem or placebo two days preoperatively and five days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* degenerative lumbar disease
* age of 18-75
* undergoing open primary one- to three-level lumbar fusion

Exclusion Criteria:

* currently use a sleep aid nightly
* diagnosed with insomnia or sleep apnea
* history of delirium with opiates or zolpidem
* allergic to opiates or zolpidem
* had previous lumbar spine surgery
* undergoing minimally invasive lumbar fusion,
* undergoing lumbar fusion for fracture, infection, tumor, or an inflammatory spondyloarthropathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Postoperative day five
  Visual analog scale (VAS) for back and leg pain; scale range: 0-10, higher scores = increased pain (worse outcome)

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Preoperative, Postoperative day three, five, as well as two weeks and six weeks
  Patient reported outcome with regard to low back pain and function; score range: 0-100%, higher scores = higher disability from low back pain (worse outcome)
Morphine Equivalents | Postoperative day one, two, three, four, five, and two weeks
  values that represent the potency of an opioid dose relative to morphine
Quality of Recovery - 40 (QoR-40) questionnaire | Preoperative, Postoperative day three, five, as well as two weeks and six weeks
  Patient Reported Outcome; score range: 40-200, higher score = greater recovery (better outcome)
Epworth Sleepiness Score (ESS) | Preoperative, Postoperative day three, five, as well as two weeks and six weeks
  Patient Reported Outcome; score range: 0-24; higher score = greater daytime sleepiness (worse outcome)
Pain Catastrophizing Scale (PCS) | Preoperative, Postoperative day three, five, as well as two weeks and six weeks
  Patient Reported Outcome; scale range: 0-24, higher score = higher pain catastrophizing (worse outcome)
Hospital Length of Stay | Postoperative two-weeks
Postoperative complications | Postoperative two-years
Visual analog scale (VAS) | preoperative, postoperative day one, three, as well as two weeks and six weeks
  Visual analog scale (VAS) for back and leg pain; scale range: 0-10, higher scores = increased pain (worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Keck Medical Center of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No